CLINICAL TRIAL: NCT05874141
Title: Comorbidities in Type 2 Diabetes Mellitus: An Observational Study in Kharga City, New Valley Governate, Egypt
Brief Title: Comorbidities in Type 2 Diabetes Mellitus
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: New Valley University (Other)
Responsible Party: Principal Investigator, Asmaa Nady Hussein, Lecturer of Internal Medicine and Clinical Hematology, New Valley University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: CODM2KNV
Record Dates: First submitted 2023-03-30; First posted 2023-05-24 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Urinalysis; Blood Cell Count

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- type 2 DM (Other)
  Interventions: Diagnostic Test: HBA1C; Diagnostic Test: Lipid profile, including total, LDL, and HDL cholesterol and Triglycerides; Diagnostic Test: Urine analysis and urinary albumin-to-creatinine ratio; Diagnostic Test: Serum creatinine and estimated glomerular filtration rate; Diagnostic Test: Complete blood count; Diagnostic Test: Thyroid-stimulating hormone; Diagnostic Test: Serum iron, TIBC, Transferrin saturation and serum ferritin if needed; Procedure: Electrocardiography (ECG); Procedure: Transthoracic echocardiography, Neck ultrasonography if needed and abdominopelvic ultrasound; Procedure: Arterial duplex ultrasound of both lower limbs; Diagnostic Test: Random blood glucose; Diagnostic Test: AST, ALT, albumin

INTERVENTIONS:
Diagnostic Test: HBA1C — blood sample on EDTA
Diagnostic Test: Lipid profile, including total, LDL, and HDL cholesterol and Triglycerides — serum sample
Diagnostic Test: Urine analysis and urinary albumin-to-creatinine ratio — Morning urine sample
Diagnostic Test: Serum creatinine and estimated glomerular filtration rate — serum sample
Diagnostic Test: Complete blood count — blood sample on EDTA
Diagnostic Test: Thyroid-stimulating hormone — serum sample
Diagnostic Test: Serum iron, TIBC, Transferrin saturation and serum ferritin if needed — serum sample
Procedure: Electrocardiography (ECG) — by electrocardiogram
Procedure: Transthoracic echocardiography, Neck ultrasonography if needed and abdominopelvic ultrasound — imaging
Procedure: Arterial duplex ultrasound of both lower limbs — imaging
Diagnostic Test: Random blood glucose — serum sample
Diagnostic Test: AST, ALT, albumin — serum sample

SUMMARY:
Type 2 diabetes mellitus (DM) has adopted a top priority as it is a disease with an increasing prevalence. The number of people living with DM has increased more than fourfold over the past 40 years to more than 460 million people today

DETAILED DESCRIPTION:
All-cause mortality rates have declined substantially in several high-income countries, including England.

A diversification in non-fatal conditions in people with DM has also been reported. This is attributable to broader, non-vascular conditions. Due to increasing longevity among people with type 2 DM with increasing and diversifying multimorbidity in them, the health needs of people with Type 2 DM are therefore likely to be broad, and complex.

Finding multimorbidity (two or more chronic conditions) is common in people with Type 2 DM and increasing, but the comorbidity profiles of people with T2DM vary substantially.

Many studies have primarily focused on identifying multimorbidity patterns in the general population.

The understanding of multimorbidity patterns and composition of specific comorbidities in people with DM, and how this varies across patient groups and during the course of the disease, is limited. Further knowledge of this could provide insight into providing more holistic and more personal approaches to clinical guideline development, care pathways, and secondary prevention.

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 2 diabetes.

Exclusion Criteria:

1. Patients with type 1 diabetes.
2. Patients with secondary diabetes.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 288 (Estimated)
Dates: Start 2023-11-15 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with hypertension | At time of inclusion in the study
Number of participants with dyslipidemia | At time of inclusion in the study
Number of participants with Diabetic kidney disease | At time of inclusion in the study
Number of participants with Coronary heart disease | At time of inclusion in the study
Number of participants with thyroid disorder | At time of inclusion in the study
Number of participants with Stroke | At time of inclusion in the study
Number of participants with Peripheral arterial disease | At time of inclusion in the study
Number of participants with Diabetic eye disease | At time of inclusion in the study
Number of participants with Peripheral neuropathy | At time of inclusion in the study
Number of participants with Liver disease | At time of inclusion in the study
Number of participants with Infections | At time of inclusion in the study
Number of participants with Cancer | At time of inclusion in the study

SECONDARY OUTCOMES:
Number of participants with controlled diabetes mellitus with correlation to the number of cormobidity | At time of inclusion in the study
Correlate the presence of each co-morbidity with the extent of diabetes control | At time of inclusion in the study

CONTACTS AND LOCATIONS:
Locations (1):
- New Valley University, Al Khārjah, Kharga Oasis, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Saeedi P, Petersohn I, Salpea P, Malanda B, Karuranga S, Unwin N, Colagiuri S, Guariguata L, Motala AA, Ogurtsova K, Shaw JE, Bright D, Williams R; IDF Diabetes Atlas Committee. Global and regional diabetes prevalence estimates for 2019 and projections for 2030 and 2045: Results from the International Diabetes Federation Diabetes Atlas, 9th edition. Diabetes Res Clin Pract. 2019 Nov;157:107843. doi: 10.1016/j.diabres.2019.107843. Epub 2019 Sep 10. PMID 31518657
- [Background] Gregg EW, Cheng YJ, Srinivasan M, Lin J, Geiss LS, Albright AL, Imperatore G. Trends in cause-specific mortality among adults with and without diagnosed diabetes in the USA: an epidemiological analysis of linked national survey and vital statistics data. Lancet. 2018 Jun 16;391(10138):2430-2440. doi: 10.1016/S0140-6736(18)30314-3. Epub 2018 May 18. PMID 29784146
- [Background] Harding JL, Shaw JE, Peeters A, Davidson S, Magliano DJ. Age-Specific Trends From 2000-2011 in All-Cause and Cause-Specific Mortality in Type 1 and Type 2 Diabetes: A Cohort Study of More Than One Million People. Diabetes Care. 2016 Jun;39(6):1018-26. doi: 10.2337/dc15-2308. Epub 2016 Apr 26. PMID 27208325
- [Background] Pearson-Stuttard J, Bennett J, Cheng YJ, Vamos EP, Cross AJ, Ezzati M, Gregg EW. Trends in predominant causes of death in individuals with and without diabetes in England from 2001 to 2018: an epidemiological analysis of linked primary care records. Lancet Diabetes Endocrinol. 2021 Mar;9(3):165-173. doi: 10.1016/S2213-8587(20)30431-9. Epub 2021 Feb 4. PMID 33549162